CLINICAL TRIAL: NCT03648255
Title: A Prospective, Observational Study to Evaluate Gastrointestinal Symptoms and Safety of an Enteral Feeding Product in Pediatric Patients With Cerebral Palsy
Brief Title: TolerUp Enteral Feeding Protocol
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA15
Record Dates: First submitted 2018-07-13; First posted 2018-08-27 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational, multi-center study will follow children with cerebral palsy who decided to switch to an enteral product that contains partially hydrolyzed protein and medium chain triglycerides as a result of clinical symptoms/diagnosis of gastrointestinal intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Fed with an enteral product that does not contain partially hydrolyzed protein and medium chain triglycerides and decided to be switched to an enteral product contains partially hydrolyzed protein and medium chain triglycerides as a result of clinical symptoms/diagnosis of gastrointestinal intolerance
* Fed by tube, using enteral tube feeding as sole source of nutrition
* A signed and dated informed consent by subject's legally acceptable representative

Exclusion Criteria:

* Chronic diseases other than cerebral palsy (e.g. diabetes mellitus, renal, liver, endocrine diseases, malignancy)
* Intestinal obstruction
* Dialysis treatment
* Requirement of artificial ventilation
* Requirement of parenteral nutrition
* Normal nutrition in addition to enteral tube feeding
* Allergy or intolerance to any ingredient of the study product
* Currently participating in another clinical or non-clinical study

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population will be composed of patients aged 1-12 and under follow-up in participating study centers in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance | Baseline to 6 months
  healthcare professional assessed

SECONDARY OUTCOMES:
Anthropometrics | Baseline to 6 months
  change in weight from baseline measurement
Care Giver Satisfaction of Enteral Product | Baseline to 6 months
  survey administered by healthcare professional

CONTACTS AND LOCATIONS:
Overall Officials: Aysugül Alptekin, MD, Study Chair — Abbott Turkey
Locations (19):
- Turkey (Türkiye) (19):
  - Çukurova University Medical Faculty, Adana
  - Hacettepe Üniversitesi University Medical Faculty, Ankara
  - Ankara Dışkapı Child Disease Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Ankara University Medical Faculty, Ankara
  - Bursa Yüksek İhtisas Research and Training Hospital, Bursa
  - Pamukkale Üniversitesi University Medical Faculty, Denizli
  - Elazığ University Medical Faculty, Elâzığ
  - Eskişehir Osmangazi University Medical Faculty, Eskişehir
  - Koç University Medical Faculty, Istanbul
  - İstanbul Kanuni Sultan Süleyman Research and Training Hospital, Istanbul
  - İstanbul Şişli Hamidiye Etfal Research and Training Hospital, Istanbul
  - İstanbul Ümraniye Research and Training Hospital, Istanbul
  - İzmir Behçet Uz Child Disease Hospital, Izmir
  - Kocaeli Üniversitesi University Medical Faculty, Kocaeli
  - Kırıkkale University Medical Faculty, Kırıkkale
  - İnönü Üniversitesi University Medical Faculty, Malatya
  - Ondokuz Mayıs University Medical Faculty, Samsun
  - Karadeniz Teknik University Medical Faculty, Trabzon

IPD SHARING:
Plan to Share IPD: Undecided